CLINICAL TRIAL: NCT06633796
Title: Pilot Experimental Study: Efficacy of Paraffin Therapy and Occupational Therapy Associated
Brief Title: Pilot Experimental Study: Efficacy of Paraffin Therapy and Occupational Therapy Associated with Robotics in Patients with Erosive Osteoarthritis
Acronym: AMADEO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Sacro Cuore Don Calabria di Negrar (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2020-60
Record Dates: First submitted 2024-10-07; First posted 2024-10-09 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Arthrosis
MeSH Terms: conditions — Osteoarthritis | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- AMADEO (Experimental): Rehabilitation treatment with occupational therapy, paraffin therapy and mobilization with robotic arm (AMADEO) of the fingers.
  Interventions: Device: AMADEO
- Standard care (Other): Rehabilitation treatment with occupational therapy and paraffin therapy.
  Interventions: Procedure: Standard of care

INTERVENTIONS:
Device: AMADEO — 304 / 5.000 The rehabilitation treatment includes 10 sessions of combined treatment of paraffin therapy, functional occupational therapy and polyarticular mobilization of the fingers with a robotic arm (Amadeo). The sessions will be scheduled 2 times a week for 5 consecutive weeks.
  Arms: AMADEO
Procedure: Standard of care — The rehabilitation treatment includes 10 sessions of combined treatment of paraffin therapy and occupational therapy for functional purposes. The sessions will be scheduled 2 times a week for 5 consecutive weeks.
  Arms: Standard care

SUMMARY:
This is a randomized, evaluator-blinded, non-profit, single-center, exploratory, medical device clinical trial aimed at evaluating the efficacy in terms of reduction of functional limitation of the combination of occupational therapy, paraffin therapy, and robotic arm mobilization compared to the center's SoC, i.e. paraffin therapy and occupational therapy.

ELIGIBILITY:
Inclusion criteria:

* Male and female patients aged between 35 and 70 years.
* Diagnosis of erosive osteoarthritis of the fingers confirmed clinically and radiologically.
* Presence of persistent functional limitation (at least 6 months) in finger flexion
* VAS value pain referred only to the hands > 5 in the week prior to enrollment in the study.
* Patients not responding to anti-inflammatory and steroid therapy used in the last 2 years.
* Patients eligible for occupational therapy and paraffin therapy.
* Signature of the Informed Consent Form for participation in the study and processing of personal data.

Exclusion criteria:

* Patients aged < 35 years and > 70 years.
* Patients with diagnosis of overlapping arthritic pathologies.
* Patients undergoing hand surgery in the 6 months prior to the evaluation.
* Patients with functional alterations to the hands due to trauma.
* Patients with cognitive or mental disorders.
* Corticosteroid use within 6 months prior to baseline.
* Patients unable to use robots with mechanical arms

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-01-25 (Actual); Primary Completion 2024-02-15 (Actual); Study Completion 2024-02-15 (Actual)

PRIMARY OUTCOMES:
VAS functionality | Baseline, 1, 3 and 6 months after treatment
  VAS scale
Dreiser index | Baseline, 1, 3 and 6 months after treatment
  Dreiser index

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Sacro Cuore Don Calabria di Negrar, Negrar, Verona, Italy